CLINICAL TRIAL: NCT00713856
Title: Comparison of Conventional and Custom With Iris Registration PRK Ablations: Assessment of Visual Function and Patient Satisfaction
Brief Title: Comparison of Conventional and Custom Photorefractive Keratectomy (PRK)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Mark Mifflin, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25339
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Custom PRK with iris registration
- 2 (Active Comparator)
  Interventions: Procedure: Conventional PRK

INTERVENTIONS:
Procedure: Custom PRK with iris registration — PRK
  Arms: 1
Procedure: Conventional PRK — PRK
  Arms: 2

SUMMARY:
The study objective is to compare the clinical outcomes using wavefront guided PRK with iris registration and conventional laser PRK using FDA-approved laser technology on the same patient.

DETAILED DESCRIPTION:
Patients undergoing bilateral PRK on the same day will have one eye randomly assigned to custom wavefront guided PRK and the fellow eye treated with conventional PRK.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed to be suitable candidates for bilateral PRK

Exclusion Criteria:

* Patients desiring monovision correction rather than bilateral distance correction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months

SECONDARY OUTCOMES:
Manifest refraction | 6 months
Wavefront aberration value | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mifflin, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, John Moran Eye Center, Salt Lake City, Utah, United States